CLINICAL TRIAL: NCT05098860
Title: Comparison of the Efficacy of Exercise, Manual Therapy and Tele-rehabilitation-Assisted Treatment on Pain, Anxiety and Quality of Life in Degenerative Cervical Diseases
Brief Title: Efficacy of Exercise, Manual Therapy and Tele-rehabilitation-Assisted Treatment on Degenerative Cervical Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Gokhan Aygul, PT,MSc, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAUMS
Record Dates: First submitted 2021-10-09; First posted 2021-10-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2021-12

CONDITIONS: Cervical Spine Disease; Neck Pain
Keywords: Pain; Anxiety; Quality of Life; Neck disability
MeSH Terms: conditions — Neck Pain; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Evaluations are made by another person who does not know about the research topic and research groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Exercise Program (Active Comparator): The home exercise program includes a general educational training program. The program includes active stretching, strengthening, and stabilization exercises of neck muscles, head and neck posture exercises as well as relaxation and diaphragmatic breathing exercises.
  Patients will be asked to do home exercises for 30-45 minutes once a day, 5 days a week for 8 weeks.
  Interventions: Other: Home Exercise Program
- Manual Therapy Combined with Home Exercise Program (Active Comparator): Manual Therapy includes soft tissue and joint mobilizations of the cervical vertebrae, scapula and thoracic vertebrae. MT will be applied to the patients 2 days a week for 8 weeks.
  The home exercise program includes active stretching, strengthening, and stabilization exercises of neck muscles, head and neck posture exercises as well as relaxation and diaphragmatic breathing exercises.
  Interventions: Other: Manual Therapy Combined with Home Exercise Program
- Tele-rehabilitation Assisted Program (Active Comparator): Tele-rehabilitation assisted program will be given in the on-line environment. During 8 weeks, regularly planned exercises will be done via online applications for 30-45 minutes 2 days a week, accompanied by a physiotherapist. These patients will apply active cervical and thoracic region mobilizations called self-mobilization. Patients will be taught active mobilization applications with the help of a towel for the cervical region, with the assistance of a foam-roller for active mobilization of the thoracic region.
  Interventions: Other: Tele-rehabilitation Assisted Program

INTERVENTIONS:
Other: Home Exercise Program — Educational training program includes active stretching, strengthening, and stabilization exercises of head and neck muscles as well as relaxation and breathing exercises.
  Arms: Home Exercise Program
Other: Manual Therapy Combined with Home Exercise Program — Manual Therapy program includes soft tissue and joint mobilizations of the cervical vertebrae, scapula and thoracic vertebrae.
  Arms: Manual Therapy Combined with Home Exercise Program
Other: Tele-rehabilitation Assisted Program — Tele-rehabilitation assisted program will be given in the on-line environment. Patients will apply active cervical and thoracic region mobilizations called self-mobilization.
  Arms: Tele-rehabilitation Assisted Program

SUMMARY:
The study aims to compare the effectiveness of soft tissue, joint mobilization, and tele-rehabilitation within the scope of Manual Therapy to the exercise program.

DETAILED DESCRIPTION:
60 subjects with cervical degenerative disease will be included in the study after a voluntary consent form is filled out. Subjects will randomly be divided into 3 groups according to the order.

Group 1:Home Exercise Program: After a general education is given to the patients, an exercise program will be taught. Patients will be asked to do home exercises for 30-45 minutes once a day, 5 days a week for 8 weeks, and fill in follow-up charts. In addition, reminder messages will be sent to these patients once a week by the physiotherapist.

Group 2: Manual Therapy Group: After a general education is given to the patients, the same exercise program will be taught. Soft tissue and joint mobilizations will be applied to the patients in this group within the scope of Manual Therapy (MT). Mobilizations of the cervical vertebrae, scapula, and thoracic vertebrae will be included. MT will be applied to the patients 2 days a week for 8 weeks.

Group 3: Tele-Rehabilitation Group: After general education, treatment will be given in the zoom environment. During the 8 weeks, regularly planned exercises will be done via Zoom for 30-45 minutes 2 days a week, accompanied by a physiotherapist. Patients will apply active cervical and thoracic region mobilizations called self-mobilization. Patients will be taught active mobilization applications with the help of a towel for the cervical region, mobilization of the thoracic region with a foam roller. Patients will apply those self-mobilization at home in front of the physiotherapist in a visual environment. Patients in this group will regularly do the same home exercises on the other days without tele-rehabilitation.

Measurement and evaluation will be done four times, as pre-treatment, post-treatment (8th week), first follow-up (12 weeks), second follow-up (6th month).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40-65
* Patients diagnosed with cervical degenerative disease
* Patients with neck pain who have had pain for at least three months
* Patients who can participate in the treatment program by following WhatsApp messages with tele-rehabilitation.

Exclusion Criteria:

* Patients with an indication for surgery for the cervical region and or a previous history of cervical surgery,
* Currently receiving treatment from another region,
* Having severe neurological loss,
* Having a primary or spinal metastatic malignancy,
* Having a vascular problem in the upper extremity,
* To be diagnosed with advanced osteoporosis,
* Being pregnant,
* Diagnosis of Diabetes Mellitus,
* Having an Inflammatory Disease (such as rheumatoid arthritis),
* Having a history of trauma,
* Those who have received physical therapy and rehabilitation for the cervical region in the last 6 months will not be included.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 8 weeks, 12 weeks and 6 months | Baseline, 8 weeks, 12 weeks, 6 months
  Visual Analog Scale will be used where patients will be asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain, at the baseline and the end of 8 weeks intervention, and at the end of 12 weeks, and 6 months from baseline.
Change from Baseline in Anxiety at 8 weeks, 12 weeks and 6 months | Baseline, 8 weeks, 12 weeks, 6 months
  Anxiety Sensitivity Index-3 will be used to evaluate the anxiety sensitivity of individuals effectively and multidimensionally. The scale is rated in a five-point Likert type and consists of a total of 18 items and is rated as 0 = very little, 4 = very much, and the total scale score ranges from 0 to 72.
Change from Baseline in Quality of Life at 8 weeks, 12 weeks and 6 months | Baseline, 8 weeks, 12 weeks, 6 months
  Nottingham Health Profile will be used to assess health-related quality of life. It is a general quality of life questionnaire that measures the individual's perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items and evaluates six dimensions related to health status: Energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). matter). Questions are answered with yes or no. Each section is scored between 0-100. 0 indicates best health, 100 indicates worst health.
Change from Baseline in Neck Disability at 8 weeks, 12 weeks and 6 months | Baseline, 8 weeks, 12 weeks, 6 months
  Neck Disability Index, consists of 10 items. Individuals included in the study will be asked to give a score between 0 (no disability) and 5 (complete disability) for each item. The total score varies between 0 (no disability) and 50 (complete disability).

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Malatya Education and Research Hospital, Malatya, Turkey (Türkiye)